CLINICAL TRIAL: NCT01531491
Title: Effects of Hypercapnia on Emergence From General Anesthesia Under Propofol: a Pilot Study
Brief Title: Effects of Hypercapnia on Emergence From General Anesthesia Under Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Junyong In, MD, Associate professor, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: J In 2011-3
Record Dates: First submitted 2012-02-06; First posted 2012-02-13 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Anesthesia, Intravenous; Anesthesia Recovery Period
Keywords: Emergence; Hypercapnia; Hypocapnia; Propofol
MeSH Terms: conditions — Hypercapnia; Hypocapnia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypercapnia group (Experimental): Respiratory rate will be 10/min and the rebreathing tube will be connected between the y-piece of corrugated tube and the tracheal tube to maintain the partial pressure of the end-tidal carbon dioxide at around 50 mmHg during emergence after propofol anesthesia.
  Interventions: Procedure: Rebreathing tube
- Hypocapnia group (Experimental): No rebreathing tube (Nothing) will be connected. Respiratory rate will be 10/min and the tidal volume will be modulated to maintain the partial pressure of the end-tidal carbon dioxide at around 30 mmHg during emergence after propofol anesthesia.
  Interventions: Procedure: No rebreathing tube (Nothing)

INTERVENTIONS:
Procedure: Rebreathing tube — 750 ml rebreathing tube will be connected between the corrugated tube and the tracheal tube of a patient. Target partial pressure of the end-tidal carbon dioxide is 50 mmHg.
  Arms: Hypercapnia group
Procedure: No rebreathing tube (Nothing) — 750 ml rebreathing tube will not be connected between the corrugated tube and the tracheal tube of a patient. Target partial pressure of the end-tidal carbon dioxide is 30 mmHg.
  Arms: Hypocapnia group

SUMMARY:
Hypercapnia derives increase of cerebral blood flow and cardiac output. It means that the rate of propofol elimination from the brain and the blood will be increased and the patient will awake more quickly. There has been no study about the effects of hypercapnia. The investigators will evaluate hypercapnia's effects on the recovery time from propofol anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA PS) I-II
* Age 20 - 60 years male and female
* Elective schedule with minor surgery under general anesthesia

Exclusion Criteria:

* Body mass index (BMI) >= 30 (kg/m2)
* Patient with pulmonary, cardiac, endocrinal, neuromuscular and neurological diseases or past history
* Patient with medication affecting on this study
* Patient with general anesthesia history within one month

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Time to open eyes under investigator's command | From cessation of propofol infusion to patient's eye opening (seconds)
  After stopping propofol infusion, every 30 seconds, the investigator (caregiver) will command the patient, "Open your eyes". When the patient opens eyes, the time will be recorded. The patients will be followed for an expected average of 10 minutes.

SECONDARY OUTCOMES:
Time to breath spontaneously | From cessation of propofol infusion to patient's spontaneous breathing (sec)
  The time from cessation of propofol infusion to patient's spontaneous breaths will be recorded. The patients will be followed for an expected average of 10 minutes.
Change of bispectral index (BIS) | From the cessation of propofol infusion to extubation, BIS and time (seconds) will be recorded.
  After stopping propofol infusion, the BIS and time (seconds) will be recorded and reviewed. These will be recorded for an expected average of 15 minutes.
Time to open mouth under investigator's command | From cessation of propofol infusion to patient's mouth opening (seconds)
  After the patient opens the eyes, every 10 seconds, the investigator command the patient, "Open your mouth.". When the patient opens mouth, the time will be recorded. The patients will be followed for an expected average of 12 minutes.
Time to extubation | From cessation of propofol infusion to extubation (sec)
  After stopping propofol infusion, When the patient breaths spontaneously with adequate tidal volume and respiratory rates, the trachea will be extubated and the time will be recorded. The patients will be followed for an expected average of 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Junyong In, M.D., Principal Investigator — Department of anesthesiology and pain medicine, Dongguk University Ilsan Hospital
Locations (1):
- Dept. of anesthesiology and pain medicine, Dongguk University Ilsan Hospital, Goyang, Kyunggido, South Korea